CLINICAL TRIAL: NCT04773977
Title: Clinical Study to Evaluate the Pharmacokinetics and Safety of IBI362 Lyophilized Powder and IBI362 Liquid Formulation in Healthy Chinese Male Subjects
Brief Title: Clinical Study of IBI362 in Healthy Chinese Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CIBI362B102
Record Dates: First submitted 2021-02-21; First posted 2021-02-26 (Actual); Last update posted 2021-07-08 (Actual); Status verified 2021-03

CONDITIONS: Overweight/Obesity
Keywords: Pharmacokinetic; Safety
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IBI362 liquid formulation (Experimental): Participants received single subcutaneous injection of IBI362 liquid formulation
  Interventions: Drug: IBI362 liquid formulation
- IBI362 lyophilized powder (Experimental): Participants received single subcutaneous injection of IBI362 lyophilized powder
  Interventions: Drug: IBI362 lyophilized powder

INTERVENTIONS:
Drug: IBI362 liquid formulation — Administered by subcutaneous injection
  Arms: IBI362 liquid formulation
Drug: IBI362 lyophilized powder — Administered by subcutaneous injection
  Arms: IBI362 lyophilized powder

SUMMARY:
This is a study to evaluate the pharmacokinetic characteristics and safety of IBI362 lyophilized powder and IBI362 liquid formulation in healthy Chinese male subjects.

DETAILED DESCRIPTION:
Pharmacokinetic；Safety

ELIGIBILITY:
Inclusion Criteria:

1. 20 years old≤ Healthy males≤45 years old
2. 19 kilograms per meter squared (kg/m²)≤Body Mass Index≤26 kg/m²
3. Willing and agreeable to commit to the duration of the study and undergo study procedures as instructed by the clinic staff

Exclusion Criteria:

1. Subjects who have previously completed or discontinued from this study, or who have used IBI362.
2. Abnormal vital signs and physical examination during the screening period;
3. Having cardiovascular, respiratory, liver, kidney, digestive, endocrine, hematologic, neurological, or muscle degenerative diseases can significantly affect drug absorption, metabolism, or elimination, or participation in the study increases risk or interferes with data interpretation.
4. Have a previous or current mental illness.
5. A family history of medullary thyroid carcinoma or multiple endocrine tumor syndrome type 2.
6. There are other factors judged by the investigators that are not suitable for inclusion in this study.

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2021-03-03 (Actual); Primary Completion 2021-03-09 (Actual); Study Completion 2021-06-17 (Actual)

PRIMARY OUTCOMES:
Evaluate the PK parameters of IBI362 in healthy Chinese male subjects | From the first dose of study drug until 8 weeks
  Peak Plasma Concentration (Cmax)
Evaluate the PK parameters of IBI362 in healthy Chinese male subjects | From the first dose of study drug until 8 weeks
  Area under the plasma concentration versus time curve (AUC)

SECONDARY OUTCOMES:
Number of Participants With Adverse Events | From the first dose of study drug until 8 weeks
  The relationship of each adverse event to the investigational product was assessed by the investigator.

CONTACTS AND LOCATIONS:
Overall Officials: Jian Li, Principal Investigator — The Sceond Affiliated Hospital of Nanchang University
Locations (1):
- The Sceond Affiliated Hospital of Nanchang University, Nanchang, China